CLINICAL TRIAL: NCT03164967
Title: A Phase IV, Multicenter, Open-label Study to Evaluate the Safety and Pharmacokinetics of BIVIGAM® in Primary Immune Deficiency Disorders in Subjects Aged 2 to 16
Brief Title: Study to Evaluate Safety and Pharmacokinetics of BIVIGAM® in Primary Immune Deficiency Subjects Aged 2 to 16
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ADMA Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 994
Record Dates: First submitted 2017-01-30; First posted 2017-05-24 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Humoral Immune Response
MeSH Terms: interventions — Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active Drug (Other): All subjects will receive Bivigam based on their prior dosing to be adjusted as clinically necessary.
  Interventions: Biological: Bivigam

INTERVENTIONS:
Biological: Bivigam

SUMMARY:
This study is part of the BIVIGAM® post marketing requirement (PMR). It is being conducted in subjects aged 2-16 with primary immune deficiency disorders associated with defects in humoral immunity to generate additional data on these populations, and more specifically safety and pharmacokinetic (PK) assessments.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/Assent
* Male or female between 2 and 16 years, inclusive, at time of Signing Informed Consent/Assent
* Have a confirmed and documented clinical diagnosis of Primary Immune Deficiency Disorder, including hypogammaglobulinemia or agammaglobulinemia.
* Have received IGIV therapy which was maintained at a steady dose (± 25% of the mean dose) for at least 3 months prior to study entry, and have maintained a trough IgG level at least 500mg/dL prior to receiving BIVIGAM®.
* Subjects and/or parents/legal guardians must be able to understand and adhere to the study visit schedule and all other protocol requirements.

Exclusion Criteria:

* Known intolerance to immunoglobulins or comparable substances (e.g. vaccination reaction).
* Known intolerance to proteins of human origin or known allergic reactions to components of the study product(s).
* Any previous randomization/participation in this clinical study must be discussed with and approved by the medical director (or designee).
* Inability or lacking motivation to participate in the study.
* Medical condition, laboratory finding, or physical exam finding (specify, e.g., vital signs outside of specific range that precludes participation. Per lab results at the Screening visit through Baseline.
* Confirmed Screening visit laboratory results ˃2.5 X ULN as defined for pediatric populations for any of the following: ALT (alanine aminotransferase/SGPT), AST (aspartate aminotransferase/SGOT), LDH (lactate dehydrogenase), BUN (blood urea nitrogen), Serum creatinine
* Has selective IgA deficiency or demonstrated antibodies to IgA.
* History of thrombotic complications of IGIV therapy or history of (deep vein thrombosis)DVT.
* Current use of daily corticosteroids (>10 mg of prednisone equivalent/day),immunosuppressants or immunomodulators are not allowed unless approved in advance by the medical monitor. Intermittent use of corticosteroids during the study is allowed if medically necessary.
* Positive diagnosis of hepatitis B or hepatitis C.
* Positive human immunodeficiency virus (HIV) test.
* Subject has had a serious bacterial infection (SBI) within the last 3 months.
* Subject has an active infection and is receiving antibiotic therapy for the treatment of this infection at the time of Screening. Note: if the subject is deemed a Screen Failure due to a nonserious active infection requiring antibiotic therapy, the subject may be rescreened 3 or 4 weeks (depending on drug administration schedule) after the initial screening.
* Subject has a history of thrombotic events (including deep vein thrombosis, myocardial infarction, cerebrovascular accident and pulmonary embolism) within 6 months before 1st IGIV dose or has preexisting risk factors for thrombotic events.
* Acquired medical condition known to cause secondary immune deficiency such as chronic lymphacitic leukemia, lymphoma or multiple lymphoma.
* Subjects with protein-losing enteropathies, hypoalbuminaemia.
* Females taking oral contraceptives.
* Pregnancy or unreliable contraceptive measures or lactation period (females of childbearing potential (female capable of becoming pregnant) only. Males capable of reproduction must agree to a double barrier method of contraception during their study participation.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Temporally Associated Adverse Events | During each infusion (During or within 1 hour, 24 hours and 72 hours of completion of an infusion)
  Incidence of adverse events (During or within 1 hour, 24 hours and 72 hours of completion of an infusion)
Number of Temporally Associated Adverse Events | Up to 72 hours of completion of an infusion
  Mean number of temporally associated per infusion
Serious Adverse Events | Up to approximately 7 months
  Incidence of serious adverse events
Related Serious Adverse Events | Up to approximately 7 months
  Incidence of related serious adverse events
Treatment Emergent Adverse Events | Up to approximately 7 months
  Incidence of treatment emergent adverse events
Related Treatment Emergent Averse Events | Within 72 hours of infusion
  Incidence of adverse events that first appear, or that worsen relative to the pre-treatment state, which occur during and within 72 hours of treatment administration
Non-treatment Emergent Adverse Events | Up to approximately 7 months
  Incidence of adverse events which do not have a causal relationship with study treatment
Temporally Associated Infusion Adverse Events | Up to approximately 7 months
  Incidence of adverse events which have a causal relationship with infusion treatment
Adverse Reactions | Up to approximately 7 months
  Number and incidence of adverse reactions plus suspected adverse reactions combined
Related Adverse Reactions | Up to approximately 7 months
  Incidence of adverse infusion related reactions
Infusion Site Reactions | Up to approximately 7 months
  Incidence reactions occuring at the infusion site
Vital Signs | Before and after each administration of study drug through study completion, up to approximately 7 months
  Change in vital signs
Temporally Associated Adverse Events Following Infusions | Up to 72 hours after each infusion through study completion, up tp approximately 7 months
  Incidence of adverse events

SECONDARY OUTCOMES:
Total IgG Trough | At each visit through study completion, up tp approximately 7 months
  Levels taken before any infusion
IgG subclasses | Prior to first and last infusion, up tp approximately 7 months
  Levels of subclasses 1- 4 before infusion
Total IgG Post | At each infusion through study completion, up tp approximately 7 months
  End of infusion level of Total IgG
Cmax | At prior to, at end of infusion, and 6 hours, 24 hours, 7 days, and 4 days, 21 days and 28 days (if still enrolled) after final infusion, up tp approximately 7 months
  Pharmacokinetic measure at 5th or 7th infusion
Tmax | At prior to, at end of infusion, and 6 hours, 24 hours, 7 days, and 4 days, 21 days and 28 days (if still enrolled) after final infusion, up tp approximately 7 months
  Pharmacokinetic measure at 5th or 7th infusion
AUC(0-ʈ) | At prior to, at end of infusion, and 6 hours, 24 hours, 7 days, and 4 days, 21 days and 28 days (if still enrolled) after final infusion, up tp approximately 7 months
  Pharmacokinetic measure at 5th or 7th infusion
AUC(0-∞) | At prior to, at end of infusion, and 6 hours, 24 hours, 7 days, and 4 days, 21 days and 28 days (if still enrolled) after infusion
  Pharmacokinetic measure at 5th or 7th infusion
Terminal phase elimination half-life (ʈ½) | At prior to, at end of infusion, and 6 hours, 24 hours, 7 days, and 4 days, 21 days and 28 days (if still enrolled) after final infusion, up tp approximately 7 months
  Pharmacokinetic measure at 5th or 7th infusion
Antibodies | At prior to, at end of infusion, and 6 hours, 24 hours, 7 days, and 4 days, 21 days and 28 days (if still enrolled) after final infusion, up tp approximately 7 months
  Levels of specific antibodies (antipneumococcal capsular polysaccharide, antihaemophilus influenza B
Infections | Up to approximately 7 months
  Number of infections of any kind, serious and non-serious
First Serious Bacterial Infection | Up to approximately 7 months
  Time to first Serious Bacterial Infections in days
Serious Bacterial Infections | Up to approximately 7 months
  Incidence of Serious Bacterial Infections
Other Infections | Up to approximately 7 months
  Incidence of infections other than Serious Bacterial Infections
Resolution of Infections | Up to approximately 7 months
  Time to resolution of Infections in days
Fever | Up to approximately 7 months
  Episodes of Fever
Missed Days | Up to approximately 7 months
  Number of days missed of school or work due to infections and treatment
Hospitalizations | Up to approximately 7 months
  Number of hospitalizations due to infections
Terminal phase elimination rate (λZ) | At prior to, at end of infusion, and 6 hours, 24 hours, 7 days, and 4 days, 21 days and 28 days (if still enrolled) after final infusion, up tp approximately 7 months
  Pharmacokinetic measure at 5th or 7th infusion

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - IMMUNOe Research Centers, Centennial, Colorado
  - Duke University Medical Center, Durham, Florida
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - USF Health, Pediatric Allergy, Immunology & Rheumatology, St. Petersburg, Florida
  - Ohio Clinical Research Associates, Mayfield Heights, Ohio
  - Oklahoma Institute of Allergy and Asthma Clinical Research, Oklahoma City, Oklahoma
  - Discovery Clinical Trials, Dallas, Texas
  - Lysosomal Rare Disorders Research & Treatment Center, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
Not yet determined